CLINICAL TRIAL: NCT04538027
Title: Effect of Duration of Symptoms on the Clinical and Functional Outcomes of Lumbar Microdiscectomy: a Randomized Controlled Trial
Brief Title: Effect of Duration of Symptoms on the Clinical and Functional Outcomes of Lumbar Microdiscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMU/Sherwan11
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Lumbar Disc Herniation
Keywords: Duration of symptoms; Outcomes; Lumbar Microdiscectomy; Oswestry disability index; Roland-Morris Questionnaire
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6 weeks (Active Comparator): Microdiscectomy was done at 6 weeks of starting symptoms
  Interventions: Procedure: Lumbar Microdiscectomy at 6 weeks of symptoms
- 3 months (Active Comparator): Microdiscectomy was done at 3 months of starting symptoms
  Interventions: Procedure: Lumbar Microdiscectomy at 3 months of symptoms
- 6 months (Active Comparator): Microdiscectomy was done at 6 months of starting symptoms
  Interventions: Procedure: Lumbar Microdiscectomy at 6 months of symptoms

INTERVENTIONS:
Procedure: Lumbar Microdiscectomy at 6 weeks of symptoms — Microscope assisted lumbar discectomy done at 6 weeks of starting symptoms
  Arms: 6 weeks
Procedure: Lumbar Microdiscectomy at 3 months of symptoms — Microscope assisted lumbar discectomy done at 3 months of starting symptoms
  Arms: 3 months
Procedure: Lumbar Microdiscectomy at 6 months of symptoms — Microscope assisted lumbar discectomy done at 6 months of starting symptoms
  Arms: 6 months

SUMMARY:
97 patients in 3 randomized groups were treated by Microdiscectomy for lumbar disc herniation; Group A was operated at 6 weeks of symptoms, Group B at 3 months and group C at 6 months. These patients were followed for 3 years for the clinical and functional outcomes.

DETAILED DESCRIPTION:
150 patients were enrolled in this study and only 97 patients were finally analyzed for primary outcomes measures of Oswestry disability index and Roland-Morris Questionnaire and secondary outcome measures of Visual analogue scale for back pain and leg pain as well as length of hospital stay and time to return for daily activities. Assessments done at different periods of 2 weeks, 3 months, 6 months, 1year, 2 years and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Disc herniation of L3-4, L4-5 or L5-S1
* MRI showed disc protrusion or extrusion with nerve root compression corresponding to clinical features.

Exclusion Criteria:

* Spondylolysis or spondylolisthesis.
* Spinal deformity like scoliosis.
* Previous spinal surgery or infection.
* Cauda equina syndrome.
* Lumbar segmental instability on dynamic radiograph: translation more than 3 mm or change in angulation more than 10 degrees
* Smoking
* Diabetes Mellitus
* Disc herniation other than levels L3-L4, L4-L5 and L5-S1
* More than single level disc hernaition.
* Body mass index 30 or more than 30
* Contained disc herniation by MRI

Ages: 19 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | Oswestry disability index was measured the functional disability at 2 weeks
  Primary outcome measure for functional disability, the higher score is better function
Roland-Morris Questionnaire | Roland-Morris Questionnaire was measured the functional disability at 2 weeks
  Primary outcome measure for functional disability, the higher score is worse function

SECONDARY OUTCOMES:
Visual analogue scale | Visual analogue scale was measured at 2 weeks
  Secondary outcome measure for back pain and leg pain, the higher score is more pain and bad results
Length of hospital stay | Measuring the days of postoperative hospital stay immediately after the surgery
  Secondary outcome measure of how many days patient remains in the hospital after operation
Return to daily activities | Measuring the time needed t return to daily activities immediately after the surgery
  Secondary outcome measure of time patient needed to return to daily activities

IPD SHARING:
Plan to Share IPD: No